CLINICAL TRIAL: NCT04739722
Title: Multitarget Stool RNA Test (ColoSense) for Colorectal Cancer Screening
Brief Title: Colorectal Cancer and Pre-Cancerous Adenoma Non-Invasive Detection Test Study
Acronym: CRC-PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geneoscopy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00045815
Record Dates: First submitted 2020-09-11; First posted 2021-02-05 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer; Advanced Adenocarcinoma; Serrated Polyp
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This phase 3 clinical trial (CRC-PREVENT) was a blinded, prospective, cross-sectional study to support a premarket approval application for a class III medical device. Subjects were recruited onto the clinical trial if they were average-risk subjects, or had a self-reported family history of CRC, aged 45 and older. All participants completed the ColoSense test, which incorporated a commercially available fecal immunochemical test (FIT), concentration of 8 RNA transcripts, and participant-reported smoking status. Stool samples were collected prior to participants completing a colonoscopy at their local endoscopy center. The ColoSense test result (positive or negative) was compared with index lesions observed on colonoscopy. The primary outcomes included ColoSense sensitivity for detecting colorectal cancer, advanced adenomas, or serrated precancerous lesions, and ColoSense specificity for all other findings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- ColoSense (Experimental): All participants were evaluated with ColoSense prior to undergoing a colonoscopy.
  Interventions: Diagnostic Test: ColoSense

INTERVENTIONS:
Diagnostic Test: ColoSense — ColoSense is intended for the qualitative detection of colorectal neoplasia-associated RNA markers and for the presence of occult hemoglobin in human stool. ColoSense is for use with the ColoSense Collection Kit, the ColoSense Test Kit, the ColoSense Software, and the following instruments: Polymedco iFOBT Analyzer; bioMérieux EMAG Nucleic Acid Extraction System; and Bio-Rad QXDx ddPCR System. ColoSense is a single-site test performed at Geneoscopy, Inc.
  A positive ColoSense result may indicate the presence of colorectal cancer (CRC), advanced adenomas (AA), or serrated precancerous lesions (SPL) and should be followed by a colonoscopy. ColoSense is indicated as a screening test for adults, 45 years of age or older, who are at typical average-risk for developing CRC. ColoSense is not a replacement for diagnostic colonoscopy or surveillance colonoscopy in high-risk individuals.

SUMMARY:
This study was a prospective analysis conducted by Geneoscopy Inc. to evaluate the ColoSense test, which is a multi-target stool RNA test for colorectal cancer screening.

DETAILED DESCRIPTION:
This phase 3 clinical trial (CRC-PREVENT) was a blinded, prospective, cross-sectional study to support a premarket approval application for a class III medical device. Subjects were recruited onto the clinical trial if they were average-risk subjects, or had a self-reported family history of CRC, aged 45 and older. All participants completed the ColoSense test, which incorporated a commercially available fecal immunochemical test (FIT), concentration of 8 RNA transcripts, and participant-reported smoking status. Stool samples were collected prior to participants completing a colonoscopy at their local endoscopy center. The ColoSense test result (positive or negative) was compared with index lesions observed on colonoscopy. The primary outcomes included ColoSense sensitivity for detecting colorectal cancer, advanced adenomas, or serrated precancerous lesions, and ColoSense specificity for all other findings.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, ≥45 years of age
* Subject is able to understand the study procedures, and is able to provide consent to participate in the study and authorizes release of relevant protected health information through reviewing and consenting to a HIPAA medical release form
* Subject is able and willing to provide stool samples within the 120 days prior to a colonoscopy procedure
* Subject is able and willing to undergo a colonoscopy after providing a stool sample

Exclusion Criteria:

* Subject had any precancerous finding on most recent colonoscopy. This does not include benign, and/or hyperplastic polyps of any size (Note: Tissue biopsies that result in no histopathology findings are acceptable)
* Subject has a history or diagnosis of colorectal cancer
* Subject has a history of aerodigestive tract cancer
* Subject has had a positive non-invasive screening diagnostic within the associated recommended intervals:

  * Fecal occult blood test or fecal immunochemical test within the previous twelve (12) months
  * FIT-DNA test within the previous 36 months
* Subject has had a colonoscopy in the previous nine (9) years
* Subject has had a prior colorectal resection for any reason other than sigmoid diverticular disease
* Indication for colonoscopy was due to overt rectal bleeding, e.g., hematochezia or melena, within the previous 30 days. (Blood on toilet paper, after wiping, does not constitute rectal bleeding)
* Subject has a diagnosis or personal history of any of the following high-risk conditions for colorectal cancer:

  * Inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease
  * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP)
  * Hereditary non-polyposis colorectal cancer syndrome (also referred to as "HNPCC" of "Lynch Syndrome")
  * Other hereditary cancer syndromes including but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Gardner's Syndrome, Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Cronkhite-Canada Syndrome, Neurofibromatosis and Familial Hyperplastic Polyposis

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14263 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Holmes, MD, Principal Investigator — Elligo Health Research
Locations (2):
- United States (2):
  - Geneoscopy, Inc., St Louis, Missouri
  - Elligo Health Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barnell EK, Wurtzler EM, La Rocca J, Fitzgerald T, Petrone J, Hao Y, Kang Y, Holmes FL, Lieberman DA. Multitarget Stool RNA Test for Colorectal Cancer Screening. JAMA. 2023 Nov 14;330(18):1760-1768. doi: 10.1001/jama.2023.22231. PMID 37870871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were engaged using an online social media platform through a decentralized recruitment effort. Interested participants completed a self-reported online survey to screen for the intended use population and to obtain socioeconomic and demographic information. Enrolled participants provided both written and oral informed consent to complete study requirements and provide medical records.
Pre-assignment Details: Of the 14,263 subjects enrolled in the CRC-PREVENT study, 8,920 completed all study requirements and 7,763 subjects were considered average-risk.
Groups:
- Enrolled Subjects: Enrolled subjects were men and women, 45 years of age or older, inclusive.
Period: Overall Study
Arm/Group | Enrolled Subjects
Started | 14263
Completed | 7763
Not Completed | 6500
Not completed — Lost to Follow-up | 5301
Not completed — Withdrawal by Subject | 42
Not completed — Non Average-risk | 1157

BASELINE CHARACTERISTICS:
Population: Subjects were men and women, 45 years of age or older, inclusive, who are at average risk of developing colorectal cancer.
Groups:
- Average Risk Subjects: Average risk subjects were required to submit a ColoSense test prior to completing a colonoscopy. Subjects were considered eligible for the primary analysis if they were 45 years or older, male or female, met eligibility criteria, and did not report a first degree relative with colorectal cancer.
Arm/Group | Average Risk Subjects
Number analyzed (Participants) | 7763
Age, Continuous [Mean (Full Range); unit: years] | 55.3 [45 to 90]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 4643
  Male | 3111
  Other | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 500
  Not Hispanic or Latino | 7121
  Unknown or Not Reported | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian / Alaskan Native | 64
  Asian | 307
  Black / African American | 821
  Native Hawaiian / Other Pacific Islander | 17
  White | 6268
  Other | 286
Region of Enrollment [Number; unit: participants]
  United States | 7763

OUTCOME MEASURES:

1. Primary Outcome: ColoSense Sensitivity for Colorectal Cancer (CRC)
Time Frame: 120 days from stool sample collection
Measure: Count of Participants; unit: Participants
Groups:
- Colorectal Cancer Subjects (Average Risk): Subjects in the average risk cohort who had a diagnosis of CRC via colonoscopy.
Arm/Group | Colorectal Cancer Subjects (Average Risk)
Number analyzed (Participants) | 27
Participants
  Positive | 25
  Negative | 2

2. Primary Outcome: ColoSense Sensitivity for Advanced Adenoma (AA)
Time Frame: 120 days from stool sample collection
Measure: Count of Participants; unit: Participants
Groups:
- Advanced Adenomas Subjects (Average Risk): Subjects in the average risk cohort who had a diagnosis of AA via colonoscopy.
Arm/Group | Advanced Adenomas Subjects (Average Risk)
Number analyzed (Participants) | 514
Participants
  Positive | 231
  Negative | 283

3. Primary Outcome: ColoSense Sensitivity for Serrated Precancerous Lesions (SPL)
Time Frame: 120 days from stool sample collection
Measure: Count of Participants; unit: Participants
Groups:
- Serrated Precancerous Lesion Subjects (Average Risk): Subjects in the average risk cohort who had a diagnosis of SPL via colonoscopy.
Arm/Group | Serrated Precancerous Lesion Subjects (Average Risk)
Number analyzed (Participants) | 98
Participants
  Positive | 22
  Negative | 76

4. Primary Outcome: ColoSense Specificity for Negative Findings
Time Frame: 120 days from stool sample collection
Measure: Count of Participants; unit: Participants
Groups:
- Negative Subjects (Average Risk): Subjects in the average risk cohort who did not have a diagnosis of CRC, AA, or SPL via colonoscopy.
Arm/Group | Negative Subjects (Average Risk)
Number analyzed (Participants) | 7124
Participants
  Positive | 1027
  Negative | 6097

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the duration of the clinical trial (From baseline to study completion, up to 120 days).
Description: Only device related adverse events were collected.
Arm/Group | Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 0/14263
Serious Adverse Events (participants affected / at risk) | 0/14263
Other Adverse Events (participants affected / at risk) | 1/14263
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=14263)
Non-serious, Anticipated, Adverse Event (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT04739722/Prot_002.pdf
  • Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT04739722/SAP_003.pdf